CLINICAL TRIAL: NCT06309693
Title: Effect of Quadratus Lumborum (QL) Block in Postoperative Pain Management Following Robotic Assisted Sacrocolpopexy
Brief Title: Postoperative Pain Management Following Robotic Assisted Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Katelyn Donaldson, MD, Fellow, Division of Urogynecology and Pelvic Reconstructive Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300011310
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse; Post Operative Pain
Keywords: minimally invasive sacrocolpopexy; quadratus lumborum block; postoperative pain; pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Pain, Postoperative | interventions — Dental Occlusion; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: The study will be a randomized control trial in which patients undergoing robotic-assisted sacrocolpopexy with concurrent robotic assisted hysterectomy or robotic assisted sacrocolpopexy after previous hysterectomy will be randomized to one of two standard of care approaches for postoperative pain management: the enhanced recovery after surgery (ERAS) protocol and the quadratus lumborum truncal nerve block. Subjects will undergo one of two standard of care approaches to postoperative pain management and be asked about their pain postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Active Comparator): The QL block will be performed by the regional anesthesia team according to their standard protocol with a uniform quantity and concentration of analgesic agent (ropivacaine 60cc). Intraoperatively, patients will undergo subcutaneous injections of lidocaine (2cc per port site) at each port site. Preoperatively, patients will only receive acetaminophen and no preoperative narcotics or neuro-modulators will be administered. Intraabdominal pressure intraoperative will be standardized among surgeons (plan for 15mm Hg for port placement, then 12 mm Hg once docked). At the conclusion of each surgery, eligible patients will receive a dose of IV ketorolac. Postoperatively, patients will be prescribed a standard regimen of NSAIDs, acetaminophen and opioids. Patients will be asked to rate their pain according to the numeric pain rating scale immediately postoperatively in the PACU and patient opioid requirements while in the PACU will be reviewed in the chart.
  Interventions: Procedure: Quadratus Lumborum (QL) Block
- Enhanced Recovery After Surgery (ERAS) Protocol (Active Comparator): The ERAS protocol is a multimodal approach to pain control while minimizing opioid medications. Subjects randomized to the ERAS arm will undergo the standard ERAS protocol of early postoperative ambulation, no bowel preparation, and the use of multimodal pain medications including acetaminophen and non-steroid anti-inflammatory drugs (NSAIDs). Intraabdominal pressure intraoperative will be standardized among surgeons (plan for 15mm Hg for port placement, then 12 mm Hg once docked). At the conclusion of each surgery, eligible patients will receive a dose of IV ketorolac. Postoperatively, patients will be prescribed a standard regimen of NSAIDs, acetaminophen and opioids. Patients will be asked to rate their pain according to the numeric pain rating scale immediately postoperatively in the PACU and patient opioid requirements while in the PACU will be reviewed in the chart.
  Interventions: Procedure: Enhanced Recovery After Surgical (ERAS) Protocol

INTERVENTIONS:
Procedure: Quadratus Lumborum (QL) Block — The standard of care QL block will be performed by the regional anesthesia team according to their standard protocol with a uniform quantity and concentration of analgesic agent. Patients will subsequently be asked about their pain postoperatively and opioid medication administration will be quantified.
  Arms: Quadratus Lumborum Block
Procedure: Enhanced Recovery After Surgical (ERAS) Protocol — Subjects randomized to the ERAS arm will undergo the standard ERAS protocol of early postoperative ambulation, no bowel preparation, and the use of multimodal pain medications including acetaminophen and non-steroid anti-inflammatory drugs (NSAIDs). Patients will subsequently be asked about their pain postoperatively and opioid medication administration will be quantified.
  Arms: Enhanced Recovery After Surgery (ERAS) Protocol

SUMMARY:
In the effort to reduce postoperative opioid use, there has been increasing interest in developing multimodal pain regimens to better manage postoperative pain while minimizing opioid use and their subsequent side effects that can be detrimental to the healing process. Standard of care approaches to better manage postoperative pain include the Enhanced Recovery After Surgery (ERAS) protocol and the use of peripheral and truncal nerve blocks. Truncal nerve blocks are widely used as an additional modality to provide longer lasting postoperative analgesia and have been adopted as part of the standard of care. The goal of this clinical trial is to compare the effects of ERAS alone versus the quadratus lumborum (QL) nerve block on the postoperative pain experience for women with pelvic organ prolapse undergoing robotic assisted sacrocolpopexy. Subjects will be randomized to the ERAS protocol or the QL block. The main questions the study aims to answer are: 1) does the QL block decrease patient reported pain scores postoperatively; and 2) does the QL block decrease the amount of opioid pain medications in the immediate postoperative period? The primary outcome measure will be median patient reported pain score in the post-anesthesia care unit (PACU) following surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare patient reported postoperative pain scores in women undergoing QL block versus ERAS protocol alone prior to minimally invasive sacrocolpopexy. Secondary aims will explore other outcomes that impact patients' overall postoperative pain experience.

Aim #1: To compare the median postoperative patient reported pain score in PACU between patients undergoing minimally invasive sacrocolpopexy, who are randomized to a preoperative QL block and the ERAS alone group.

Aim #2: To compare the maximum postoperative patient reported pain score in PACU between patients undergoing minimally invasive sacrocolpopexy, who are randomized to a preoperative QL block and the ERAS alone group.

Aim #3: To compare the total oral morphine equivalents (OME) in PACU between patients undergoing minimally invasive sacrocolpopexy, who are randomized to a preoperative QL block and the ERAS alone group.

Aim #4: To compare the rates of postoperative nausea and vomiting (PONV between patients in the QL block and ERAS alone groups undergoing minimally invasive sacrocolpopexy.

Aim #5: To compare the rates of overnight admission between patients in the QL block and ERAS alone groups undergoing minimally invasive sacrocolpopexy.

Aim #6: To compare the total time in the PACU between patients in the QL block and ERAS alone groups undergoing minimally invasive sacrocolpopexy.

Aim #7: To compare the rates of initial active voiding trial failures between patients in the QL block and ERAS alone groups undergoing minimally invasive sacrocolpopexy.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing robotic-assisted sacrocolpopexy with concurrent robotic assisted supracervical or total laparoscopic hysterectomy or robotic assisted sacrocolpopexy after previous hysterectomy
2. Age 18 years old or greater
3. Fluency and literacy in English
4. Capacity to provide consent

Exclusion Criteria:

1. Lack fluency and literacy in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Median postoperative patient reported pain score in post-anesthesia recovery unit (PACU) | Immediate postoperative period while patient is in the PACU
  Patients will be asked to rate their pain according to the numeric pain rating scale (0-10) by the nursing staff postoperatively at regular intervals in the PACU and the median score will be calculated.

SECONDARY OUTCOMES:
Maximum postoperative patient reported pain score in PACU | Immediate postoperative period while patient is in the PACU
  Patients will be asked to rate their pain according to the numeric pain rating scale (0-10) by the nursing staff postoperatively at regular intervals in the PACU and the maximum score will be identified.
Total oral morphine equivalents (OME) required in PACU Total oral morphine equivalents (OME) required in post-anesthesia recovery unit | Immediate postoperative period while patient is in the PACU
  The total quantities of opioid pain medications will be identified on patient chart review and calculated into total OME.
Rates of postoperative nausea and vomiting (PONV) in PACU | Immediate postoperative period while patient is in PACU
  Rates of PONV will be determine by administration of anti-emetic medication in PACU or documentation of PONV in notes.
Rates of overnight admission | Day of surgery
  Chart review will be performed to identify patients admitted postoperatively excluding planned admissions.
Total time spent in PACU | Immediate postoperative period while patient is in the PACU
  The total time spent in PACU will be calculated based on chart review.
Rates of initial active voiding trial failures | Immediate postoperative period while patient is in the post-anesthesia recovery unit
  The rates of initial voiding trial failures will be calculated based on chart review.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Mavarez AC, Hendrix JM, Ahmed AA. Transabdominal Plane Block. 2023 Nov 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560527/ PMID 32809362
- [Background] Dhanjal ST, Tonder S. Quadratus Lumborum Block. 2023 Aug 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537212/ PMID 30725897
- [Background] El Hachem L, Small E, Chung P, Moshier EL, Friedman K, Fenske SS, Gretz HF 3rd. Randomized controlled double-blind trial of transversus abdominis plane block versus trocar site infiltration in gynecologic laparoscopy. Am J Obstet Gynecol. 2015 Feb;212(2):182.e1-9. doi: 10.1016/j.ajog.2014.07.049. Epub 2014 Aug 1. PMID 25088860
- [Background] Hotujec BT, Spencer RJ, Donnelly MJ, Bruggink SM, Rose SL, Al-Niaimi A, Chappell R, Stewart SL, Kushner DM. Transversus abdominis plane block in robotic gynecologic oncology: a randomized, placebo-controlled trial. Gynecol Oncol. 2015 Mar;136(3):460-5. doi: 10.1016/j.ygyno.2014.11.013. Epub 2014 Nov 20. PMID 25462201
- [Background] Zoorob D, Tsolakian I, Shuffle E, Perring P, Maxwell R. Addition of Transversus Abdominis Plane Block to Conventional Pain Regimens in Robotic Sacrocolpopexy Procedures-A Pilot Randomized Controlled Trial (SACROTAP). Urogynecology (Phila). 2023 Feb 1;29(2):139-143. doi: 10.1097/SPV.0000000000001287. PMID 36735426
- [Background] Fujimoto H, Irie T, Mihara T, Mizuno Y, Nomura T, Goto T. Effect of posterior quadratus lumborum blockade on the quality of recovery after major gynaecological laparoscopic surgery: A randomized controlled trial. Anaesth Intensive Care. 2019 Mar;47(2):146-151. doi: 10.1177/0310057X19838765. Epub 2019 May 15. PMID 31090440
- [Background] Hansen C, Dam M, Nielsen MV, Tanggaard KB, Poulsen TD, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block for total laparoscopic hysterectomy: a double-blind, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2021 Jan;46(1):25-30. doi: 10.1136/rapm-2020-101931. Epub 2020 Oct 20. PMID 33082286
- [Background] Jiang W, Wang M, Wang X, Jin S, Zhang M, Zhang L, Zhang Y, Wu Y. Effects of Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block on Postoperative Opioid Consumption in Total Laparoscopic Hysterectomy: A Randomized Controlled Clinical Trial. Pain Ther. 2023 Jun;12(3):811-824. doi: 10.1007/s40122-023-00505-1. Epub 2023 Apr 13. PMID 37052813
- [Background] Jadon A, Ahmad A, Sahoo RK, Sinha N, Chakraborty S, Bakshi A. Efficacy of transmuscular quadratus lumborum block in the multimodal regimen for postoperative analgesia after total laparoscopic hysterectomy: A prospective randomised double-blinded study. Indian J Anaesth. 2021 May;65(5):362-368. doi: 10.4103/ija.IJA_1258_20. Epub 2021 May 20. PMID 34211193
- [Background] Scheib SA, Thomassee M, Kenner JL. Enhanced Recovery after Surgery in Gynecology: A Review of the Literature. J Minim Invasive Gynecol. 2019 Feb;26(2):327-343. doi: 10.1016/j.jmig.2018.12.010. Epub 2018 Dec 20. PMID 30580100